CLINICAL TRIAL: NCT00659113
Title: A Phase II Trial of a TS-1/Cisplatin Based Definitive Chemoradiotherapy for Resectable Esophageal Cancer
Brief Title: S-1, Cisplatin, and Radiation Therapy in Treating Patients With Stage IIA, Stage III, or Stage IVA Esophageal Cancer That Can Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593402; YONSEI-4-2007-0342
Record Dates: First submitted 2008-04-15; First posted 2008-04-16 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2008-12

CONDITIONS: Esophageal Cancer
Keywords: stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Endoscopic Mucosal Resection

INTERVENTIONS:
Drug: cisplatin
Drug: tegafur-gimeracil-oteracil potassium
Other: cytology specimen collection procedure
Procedure: endoscopic biopsy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as S-1 and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy together with more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving S-1 and cisplatin together with radiation therapy works in treating patients with stage IIA, stage III, or stage IVA esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate response rate in patients with stage IIA-IVA resectable esophageal cancer treated with chemoradiotherapy comprising S-1, cisplatin, and radiotherapy.

Secondary

* To evaluate overall survival of these patients.
* To evaluate progression-free survival of these patients.
* To evaluate toxicity in these patients.
* To correlate initial squamous cell carcinoma antigen and C-reactive protein with response and survival in these patients.

OUTLINE: Patients receive oral S-1 twice weekly, cisplatin IV over 2 hours on day 1, and undergo radiotherapy 5 days a week in weeks 1 and 2. Treatment repeats every 3 weeks for 2 courses.

Tumor tissue samples are collected by esophagoscopy with biopsy and brushings for analysis of initial squamous cell carcinoma antigen and C-reactive protein correlation with response and survival.

After completion of study treatment, patients are followed for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the esophagus

  * Stage IIA-IVA disease
  * Resectable disease
* Measurable disease, defined as at least 1 measurable lesion by RECIST criteria
* No known brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* ANC ≥ 1,500/uL
* Hemoglobin ≥ 9.0 g/dL (transfusion correction allowed)
* Platelets ≥ 100,000/uL
* Creatinine < 1.5 mg/dL
* Total bilirubin < 2 times upper limit of normal (ULN)
* ALT/AST < 3 times ULN
* Fertile patients must use effective contraception
* Not pregnant or nursing
* Able to take oral medication
* No active peptic ulcer disease
* No known hypersensitivity to study drugs
* No serious uncontrolled systemic intercurrent illness, including the following:

  * Poorly controlled diabetes
  * Active infection
* No history of significant neurological or mental disorder, including seizures or dementia
* No malignancy within the past 5 years, except carcinoma in situ of the cervix, or nonmelanomatous carcinoma of the skin
* No active cardiac disease uncontrolled by therapy
* No myocardial infarction within the past 12 months
* No interstitial lung disease or extended fibrosis of lung

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for esophageal cancer
* No prior surgical procedure affecting absorption
* No concurrent flucytosine or other fluoropyrimidine-group anticancer drugs
* No concurrent systemic chemotherapy, investigational drug, or radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-03

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Overall survival
Progression-free survival
Toxicity
Initial squamous cell carcinoma antigen and C-reactive protein correlation with response and survival

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hang Kim, MD, Study Chair — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea